CLINICAL TRIAL: NCT02756702
Title: Prospective Observational 5 Year Follow-up on a Consecutive Cohort of 70 Primary Total Knee Arthroplasty (TKA) Cases Treated With All-polyethylene Tibia (APT) Components of the Posterior-stabilized VEGA System PS
Brief Title: All Polyethylene Tibia-VEGA Kiel
Acronym: APT-VEGA_KI
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Collaborators: Frictionless GmbH, Kiel (Unknown)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1527
Record Dates: First submitted 2016-04-27; First posted 2016-04-29 (Estimated); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Degenerative Osteoarthritis; Rheumatoid Arthritis; Post-traumatic; Arthrosis; Other Instability, Knee; Stiffness of Knee, Not Elsewhere Classified; Deformity of Knee Joint
Keywords: TKA; TKR; All-Poly; posterior stabilized
MeSH Terms: conditions — Joint Diseases; Arthritis, Rheumatoid; Osteoarthritis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All-Poly: All-polyethylene tibia VEGA System® PS - A posterior stabilized total knee arthroplasty (TKA) system using solely all-polyethylene tibia components
  Interventions: Device: All-Poly

INTERVENTIONS:
Device: All-Poly — Implantation of the VEGA PS using all-polyethylene tibia components
  Other Names: Total Knee Replacement

SUMMARY:
Obligatory Post-Marketing Clinical Follow-up (PMCF) as part of the post marketing surveillance plan for the product under investigation For this PMCF only CE-marked medical devices will be used within their intended purpose and no additional invasive or other stressful examinations are to be carried out (acc. to MPG §23b).

DETAILED DESCRIPTION:
This non-interventional clinical study (NIS) is conducted to clinically confirm the safety and performance of the Aesculap® APT VEGA System® PS components under routine conditions. The VEGA System® PS is an established TKA design, and there is a long-lasting experience in the use of PE for TKA in general and for APT components in particular; thus a NIS is thought to be sufficient to give the required confirmation. For this NIS only CE-marked medical devices will be used within their intended purpose and no additional invasive or other stressful examinations are to be carried out (acc. to MPG §23b). As part of the post marketing surveillance plan an obligatory Post-Marketing Clinical Follow-up (PMCF) is required for the product under investigation.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring primary TKA because of severe knee joint conditions that cannot be treated through other therapies;
* degenerative osteoarthritis;
* rheumatoid arthritis;
* posttraumatic arthritis;
* symptomatic knee instability;
* knee stiffness or deformation of the knee joint;
* Age ≥ 18 years;
* Patient signed informed consent

Exclusion Criteria:

* Age younger than 18 years
* Any prior joint replacement at the index knee
* Unable or unwilling to return for postoperative follow-up
* Patient did not sign informed consent
* Joint conditions that can be treated by reconstructive surgery (e.g. osteotomy)
* Acute or chronic infections near the joint, or systemic infections
* Secondary diseases that could influence joint implant functionality
* Systemic diseases and metabolic disorders
* Severe osteoporosis or osteomalacia
* Severely damaged bone structures that could prevent stable implantation of implant components
* Bone tumors in the region of implant fixation
* Bone malformations, axial misalignments or other bone conditions that rule out implantation of a prosthetic joint
* Expected overload on the joint implant, especially due to high patient weight or intense physical strain and activity
* Dependency on pharmaceutical drugs, drug abuse, or alcoholism
* Fever, infection or inflammation (systemic or local)
* Pregnancy
* Mental illness
* Severe osteopenia (or any other medical or surgical finding) that would preclude any benefit from the implants
* Combination with implant components from other manufacturers
* Inadequate patient compliance
* Foreign body sensitivity to the implant materials
* All cases not listed under indications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2022-10-06 (Actual)

PRIMARY OUTCOMES:
Revision Rate | 5 years
  The objective of the study is to collect clinical midterm outcome information on the product under investigation when used in routine clinical practice.

SECONDARY OUTCOMES:
Complication/Adverse Event rate | 5 years
  Cumulative Number of Complications / Adverse Events of any reason over the period of follow-up
KOOS (Knee Osteoarthritis Outcome Score) | 5 years
  Changes of the total Knee injury and Osteoarthritis Outcome Score (KOOS) from the preoperative baseline to the 5-year postoperative
KSS (Knee Society Score) | 5 years
  Changes of the Knee Society Score (KSS) with its Knee and Functional Score (KS and FS) from the preoperative baseline to the 5-year postoperative assessment
SF-12® Health Survey (SF-12) | 5 years
  Changes of the total SF-12® Health Survey (SF-12) components Physical Component Summary (PCS-12) and Mental Component Summary (MCS-12) from the preoperative baseline to the 5-year postoperative assessment
Change of anterior knee pain over follow-up period | 5 years
  Changes of anterior knee pain according to the Waters and Bentley rating system from the preoperative baseline to the 5-year postoperative assessment

CONTACTS AND LOCATIONS:
Overall Officials: Ludger Gerdesmeyer, Professor, Principal Investigator — orthopedics
Locations (1):
- MEDBALTIC GmbH c/o Mare Klinikum, Kiel, Germany

IPD SHARING:
Plan to Share IPD: No